CLINICAL TRIAL: NCT06319794
Title: A Randomized Phase 2 Proof-of-Concept Study to Evaluate the Efficacy and Safety of Topical Bimiralisib Application in Participants Suffering From Actinic Keratosis on the Face and/or Scalp and/or Back of Hands Over a 2 and 4-week Treatment Period
Brief Title: Study on the Safety and Efficacy of Bimiralisib Gel in Participants Suffering From Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TORQUR (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQR-BTOP-101
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimiralisib - 2 weeks treatment (Experimental): Topical bimiralisib for 2 weeks
  Interventions: Drug: Bimiralisib
- Bimiralisib - 4 weeks treatment (Experimental): Topical bimiralisib for 4 weeks
  Interventions: Drug: Bimiralisib

INTERVENTIONS:
Drug: Bimiralisib — Participants will be instructed to self-apply topical bimiralisib gel on the treatment area once daily for 2 weeks
  Arms: Bimiralisib - 2 weeks treatment
Drug: Bimiralisib — Participants will be instructed to self-apply topical bimiralisib gel on the treatment area once daily for 4 weeks
  Arms: Bimiralisib - 4 weeks treatment

SUMMARY:
The aim of the study is to evaluate efficacy and safety of bimiralisib gel treatment for treatment of actinic keratosis (AK) on the face and/or scalp and/or back of hands

DETAILED DESCRIPTION:
This is a multi-center, randomized, open label, parallel group study. The study products will be applied to the target lesions for a duration of 2 or 4 weeks of treatment.

The study consists of the following periods:

* Screening (up to 30 days)
* Treatment (2 or 4 weeks)
* Follow-Up (4 weeks)

Participants will be randomized to one of two groups (1:1):

* Arm A: Topical bimiralisib gel treatment for 2 weeks
* Arm B: Topical bimiralisib gel treatment for 4 weeks

ELIGIBILITY:
Key Inclusion Criteria:

* Must be of at least 50 years of age, at the time of signing the informed consent.
* Have a clinical diagnosis of stable, clinically typical actinic keratosis.
* Have at least 3 actinic keratosis lesions contained within contiguous treatment regions of face and/or scalp and/or back of hands.
* Must agree not to use any product on the treatment area during the entire course of study except for Investigator-approved cleanser, sunscreen, wash, and non-medicated makeup.
* Must be willing to comply with sun avoidance measures for all exposed areas including use of Investigator-approved sunscreen and/or hats, have limited sun exposure time, and have no tanning bed use.
* Must be in good general health (ECOG 0-1)
* Participants of reproductive potential must agree to use double effective contraception from screening until 90 days after discontinuing study treatment.
* Female participants who had a menstrual cycle within 2 years prior to screening must have a negative serum pregnancy test at screening and a negative urine pregnancy test on their first treatment day.
* Must be capable of giving signed informed consent

Key Exclusion Criteria:

* Known or suspected hypersensitivity to any of the excipients of bimiralisib gel.
* Clinically atypical and/or rapidly changing actinic keratosis lesions in the treatment area.
* Clinical evidence of severe, uncontrolled autoimmune, cardiovascular, gastrointestinal, hematological, hepatic, neurologic, pulmonary or renal disease.
* Participation in any clinical research study within 30 days of the Baseline Visit.
* Cosmetic or therapeutic procedures (e.g. laser, peeling, photodynamic therapy, cryotherapy) within 4 weeks of the Baseline visit and within 2 cm of the selected treatment area.
* Use of sun lamps, tanning beds, and tanning booths during the 4 weeks prior to the Baseline Visit or planned use during the study.
* Use of any retinoids within 90 days of the Baseline Visit, or glucocorticosteroids, methotrexate or other anti-metabolites or nicotinamide within 28 days of the Baseline Visit.
* Any systemic cancer therapy or diagnosis within 6 months of the Baseline Visit.
* Any other malignancy within 5 years prior to Screening except basal or squamous cell carcinoma not in the treatment area that were treated with curative intent and are without recurrence.
* Other significant uncontrolled or unstable medical diseases or conditions that, in the opinion of the Investigator, would expose the participant to unacceptable risk by study participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in AK lesions as measured by achieving an Investigator Global Assessment (IGA) score of 0 or 1 | Baseline, Day 43 (Treatment Arm A), Day 57 (Treatment Arm B)
  Improvement from baseline in AK lesions as measured by achieving an Investigator Global Assessment (IGA) score of 0 or 1 (on a 0-4 scale where 0 is complete clearance and 4 is no improvement)

SECONDARY OUTCOMES:
Proportion of participants with partial or complete clearance of AK lesions at the End of Treatment Visit (Week 2 or 4 depending on treatment arms) | Day 15 (Treatment Arm A), Day 29 (Treatment Arm B)
  Proportion of participants with partial (75% reduction in lesions) or complete clearance of AK lesions at the End of Treatment Visit (Week 2 or 4 depending on treatment arm)
Incidence of Treatment-Emergent Adverse Events | From first application of bimiralisib until 28 days after the last application
  Safety endpoint assessed by treatment-emergent adverse events (including laboratory adverse events and vital signs)
Incidence of local skin reactions | From first application of bimiralisib until 28 days after the last application
  Tolerability endpoint assessed by Investigator for specific local skin reactions using 4-point clinical scales for irritation, stinging/burning and pruritus.
  Scales from 0 (no signs) to 3 (severe)

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Hospital Basel / Department of Dermatology, Basel
  - CHUV centre hospitalier universitaire vaudois / Department of Dermatology and Venereology, Lausanne

IPD SHARING:
Plan to Share IPD: No